CLINICAL TRIAL: NCT06796478
Title: Effects of Tailored Egoscue Exercises on Pain, Functional Performance and Sleep Quality in Patients With Lumbar Radiculopathy
Brief Title: Tailored Egoscue Exercises in Patients With Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0213NamraSarwar
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Radiculopathy
Keywords: egoscue excercises; lumbar radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 10 minutes of heat therapy and 30 minutes of tailored Egoscue excercises
  Interventions: Other: Tailored Egoscue Excercises
- Group B (Active Comparator): 10 minutes of heat therapy & core stabilization exercises employed for 30 minutes.
  Interventions: Other: Core stabilization excercises

INTERVENTIONS:
Other: Tailored Egoscue Excercises — A. Elbow curls on the wall with abduction B. Elbow curls on the wall with adduction C. Overhead extension D. Open Up arm and chest E. Upper spinal twist. F. Spinal Twist G. Pelvic tilts H. Static back alone and static back with breathing I. Static wall. J. Air Bench Abdominal contraction in the static back position. K. Resisted Abduction L. Abductor press M. Supine groin progression
  Arms: Group A
Other: Core stabilization excercises — A. Cat Pose & Camel pose B. Pelvic tilt C. Hip flexor stretches D. Hamstring stretches E. Piriformis stretch F. Prone on elbow
  Arms: Group B

SUMMARY:
Lumbar radiculopathy (LR), commonly sciatica, is characterized by inflammation of the lower back's nerve roots. It is typically caused by sensory disruptions that arise from the lumbar spine and extend downward below the knee. LR is marked by alterations in motor and sensory functions, such as Radicular discomfort,functional performance paresthesia, or tingling in the lower limb.

This research aims to explore the Effects of Tailored Egoscue Exercises on Pain, Functional Performance and Sleep Quality in Patients with Lumbar Radiculopathy

DETAILED DESCRIPTION:
The study was a randomized controlled trial, total 54 patients were recruited from Rayan Medical Center, Gujrat by using probability convenience sampling technique and assigned into two equal groups .27 patients in Group A (Experimental group) did Egoscue exercises while Group B (Control group) was provided with routine rehabilitation. In this study, age group between 45 to 65 pre-diagnosed with lumbar radiculopathy by a neurophysician was included. Lasègue's test , Bragard's test and Slump test was performed as a screening tool in the study. Exercises was performed for 40 minutes per day on 3 alternate days per week for 6 weeks.Group A (Experimental Group) included 10 minutes of heat therapy and 30 minutes of Egoscue training while at Group B (Control Group) 10 minutes of heat therapy, gentle stretches & core stabilization exercises for 30 minutes was performed. Patients was assessed at three levels pre (at baseline), mid (after 3 weeks) and post level(after 6 weeks) . Assessment tool was a Numerical pain rating Scale, Rolland-Morris Disability Questionnaire & Insomnia Severity Index (ISI) to assess the outcome variable

ELIGIBILITY:
Inclusion Criteria:

* Age 45-65 years
* Both male and female
* Lumbar disc herniation /lumbar radiculopathy secondary to L4/L5 and L5/S1
* Patients diagnosed with lumbar radiculopathy by neuro physician
* Positive Lasègue's test(SLRT): Positive if pain occurs when the hip is flexed at 30 and 60 or 70 degrees from horizontal.
* Positive Bragrd's sign: Applying ankle dorsiflexion after the straight leg raise (SLR) with the knee extended causes pain.
* Positive Slump test: positive if symptoms are increased in the slumped position and decreased as the patient moves out of neck flexion

Exclusion Criteria:

* Received treatment for LBP in the past 6 months
* Practiced any kind of exercise or sports activity during the last 6 months
* spinal tumors
* infections
* pregnancy
* neoplasm

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS): | 6weeks
  The NPRS is commonly used for assessing the intensity of pain, requiring patients to indicate their pain severity by choosing a number on a scale ranging from 0 to 10. This implies that a Numeric Rating Scale (NRS) score within the 1-5 range indicates a mild disruption in functioning, scores of 6 and 7 denote moderate interference and a score within the 8-10 range signifies severe interference with functionality. The pain scale spans from zero, indicating no pain, to ten, signifying the utmost agony. Reliable test-retest consistency has been evidenced through NPRS, with correlation coefficients of 0.96 and 0.95, respectively.
The Roland Morris Disability Questionnaire (RMDQ) | 6weeks
  It was employed to assess patients' functional limitations. The RMQ, a patient-reported outcome measure consisting of 24 items, assesses disability related to pain arising from lower back pain. Each item is assigned a score of 0 if left unanswered or 1 if affirmed, resulting in a total RMQ score that ranges from 0 to 24. Elevated scores indicate greater levels of pain-related disability. Therefore, a higher numerical value is indicative of more pronounced lumbago severity. Upon examination of the 24 items, it becomes apparent that they encompass a diverse range of aspects. Some items appear linked to the physical facets of quality of life (QOL), while others likely capture different dimensions of QOL. The RMDQ has demonstrated a high level of internal consistency reliability (Cronbach's alpha of 0.87) and test-retest reliability (ICC of 0.9). A change of 2-3 points (8-12%) is considered clinically significant
Insomnia Severity Index (ISI) questionnaire | 6weeks
  A self-reported questionnaire called the Insomnia Severity Index (ISI) is used to assess how well people slept over the previous month.
  The seven-item questionnaire, which is a quick screening tool for insomnia, asks participants to use a Likert-style scale to score the kind and severity of their sleep issues. Questions about subjective aspects of the respondent's sleep include how severe symptoms are, how satisfied the respondent is with their sleep patterns, how much insomnia interferes with day-to-day functioning, how obvious they believe their insomnia is to others, and how much distress the sleep issue causes them overall. Management The short scale is a pencil-and-paper self-report measure that takes only roughly five minutes to complete.
  It found item-total correlations that were very varied, ranging from 36 to 54, and had an internal consistency of a =.74. Likert-type scales are used by respondents to score each component of the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Rayan Medical center, Gujrat, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No